CLINICAL TRIAL: NCT03068195
Title: Efficacy and Safety of Microwave Ablation in BosniakⅠ~ⅡF Cystic Renal Lesions: Clinical Outcomes of a Randomised Controlled Trial
Brief Title: Efficacy and Safety of Microwave Ablation in BosniakⅠ~ⅡF Cystic Renal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-20161017
Record Dates: First submitted 2017-02-18; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Kidney Diseases,Cystic
Keywords: laparoscopy; microwave; ablation technique
MeSH Terms: conditions — Kidney Diseases, Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- laparoscopic microwave ablation (Experimental): laparoscopic microwave ablation will be performed before the renal cysts are decorticated
  Interventions: Procedure: microwave ablation
- percutaneous microwave ablation (Experimental): percutaneous microwave ablation will be performed to treat the renal cysts without decorticating.
  Interventions: Procedure: microwave ablation
- laparoscopic decortication (Active Comparator): conventional laparoscopic decortication will be performed to treat the renal cysts.
  Interventions: Procedure: laparoscopic decortication

INTERVENTIONS:
Procedure: microwave ablation — KY2000 microwave ablation system was used in the experimental group. A power output of 60 W for 1-3 min for 1-3 cycles to treat the renal cysts according to the cysts size and classification.Percutaneous microwave ablation will be performed under the guidance of ultrasound while the laparoscopic microwave ablation will be performed under direct vision
  Arms: laparoscopic microwave ablation; percutaneous microwave ablation
Procedure: laparoscopic decortication — conventional laparoscopic decortication will be performed to treat the renal cysts
  Arms: laparoscopic decortication

SUMMARY:
The purpose of this study is to determine whether microwave ablation is more effective in the treatment of simple renal cysts than conventional laparoscopic decortication.

DETAILED DESCRIPTION:
Background: Simple renal cysts are the most common renal masses, and occur in half of all patients older than 50 years.They are usually asymptomatic and benign, asymptomatic and discovered incidentally. However, over time, these simple cysts can enlarge, become symptomatic and develop complications, requiring intervention.They can be managed by a variety of surgical and percutaneous methods, including percutaneous aspiration (with or without injection of a sclerosing agent), endoscopic marsupialization or excision, open surgery and laparoscopic cyst excision.Percutaneous aspiration and sclerotherapy have been described as safe and effective methods of managing symptomatic simple renal cysts without the cost and morbidity associated with conventional surgery and laparoscopy.However, laparoscopic decortications and simple aspiration is associated with a high recurrence rate because the cyst wall epithelium is responsible for active liquid production.

Purpose:To determine whether microwave ablation is more effective in the treatment of simple renal cysts than conventional laparoscopic decortication.

Method:

ELIGIBILITY:
Inclusion Criteria:

* patients with sporadic, unilateral, newly diagnosed Bosniak Ⅰ, Ⅱ and ⅡF renal cyst
* patients agreeable to participate in this long-term follow-up study
* patients with normal contralateral renal function (differential renal function of >40% as determined by radionuclide scintigraphy)

Exclusion Criteria:

* patients' aged >80 years
* patients not able to tolerate the microwave ablation procedure
* patients with previous renal surgery or history of any inflammatory conditions of the operative kidney
* patients with the renal cyst involving urinary collecting system
* patients with other renal diseases,(including kidney stone, glomerular nephritis, etc.) which might affect the renal function of the operative kidney

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
local recurrence | 12 months postoperatively

SECONDARY OUTCOMES:
postoperative complications | postoperative，up to 30 days
operative time | during operation
Hospital stay time | time from the date of admission until the date of discharge, up to 2 weeks
quality of life assessed by quality of life questionnaire | postoperative，up to 6 months
change from baseline glomerular filtration rate (GFR) of the affected kidney, 12 months minus baseline | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yiran Huang, Study Director — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Yonghui Chen, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No